CLINICAL TRIAL: NCT01361347
Title: Phase 4 Study: Milk Oral Immunotherapy for Cow's Milk Allergy in School-aged Children
Brief Title: Safety of Oral Immunotherapy for Cow's Milk Allergy in School-aged Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Marita Paassilta, MD, PhD, Paediatric Allergist, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PaassiltaM
Record Dates: First submitted 2011-02-24; First posted 2011-05-26 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Milk Allergy; Anaphylaxis
Keywords: milk allergy; desensitization; anaphylaxis; school-age
MeSH Terms: conditions — Milk Hypersensitivity; Anaphylaxis | interventions — Milk; Desensitization, Psychologic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): rice/soy/oat "milk"drink, masked
  Interventions: Dietary Supplement: milk
- milk (Experimental): cow's milk
  Interventions: Dietary Supplement: milk

INTERVENTIONS:
Dietary Supplement: milk — milk for milk allergic children (1:25 dilution, whole milk)
  Other Names: milk allergy; desensitization

SUMMARY:
The purpose of this study is to study the number of Participants with Adverse Events as a Measure of Safety and Tolerability.

DETAILED DESCRIPTION:
Eligibility criteria:

Age 6 - 16 yrs

* IgE-mediated milk allergy
* and milk provocation within 3 months prior to or an documented accidental milk contact with clear immediate symptoms

Outcome measures:

* number of patients with successful desensitization (195 - 200 ml milk per day)
* number of patients with adverse events

ELIGIBILITY:
Inclusion Criteria:

* IgE-mediated milk allergy
* An immediately positive challenge test result to milk prior to inclusion

Exclusion Criteria:

* Not willing to participate

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2008-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 12 months

SECONDARY OUTCOMES:
Number of participants drinking 2 dl/day of milk (success in desensitization) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marita Paassilta, MD, PhD, Principal Investigator — Consultant Pediatric Allergist
Locations (1):
- Tampere University Hospital, Allergy Centre, Tampere, Finland